CLINICAL TRIAL: NCT06496594
Title: Ultrasonic Scaler VS Erythritol for Peri-implant Maintenance of Loaded Implants With Crowns Made by Different Materials: 12-months Randomized Clinical Trial
Brief Title: Ultrasonic Scaler VS Erythritol for Peri-implant Maintenance of Loaded Implants With Crowns Made by Different Materials
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Andrea Scribante, Associate Professor, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-CROWNSHYGIENE
Record Dates: First submitted 2024-07-03; First posted 2024-07-11 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Peri-implant Mucositis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Erythritol group (Experimental)
  Interventions: Other: Erythritol prophylactic powders
- Ultrasonic scaler (Active Comparator)
  Interventions: Other: Ultrasonic scaler with peek inserts

INTERVENTIONS:
Other: Erythritol prophylactic powders — erythritol with particle size of ~14 µm will be used for 5 seconds (AIRFLOW® PLUS EMS)
  Arms: Erythritol group
Other: Ultrasonic scaler with peek inserts — ultrasonic scaler, a piezoelectric handpiece with peek inserts (Mini Piezon EMS; PI, EMS) will be used.
  Arms: Ultrasonic scaler

SUMMARY:
The aim of the study is to assess the effect of a 12-month peri-implant protocol with erythritol orultrasonic scaler with peek inserts for dental implants with crowns made by different materials .

Patients will be randomly divided into two groups:

Erythritol group: erythritol with a particle size of ~14 µm will be used for 5 seconds (AIRFLOW® PLUS EMS) Ultrasonic scaler group: a piezoelectric handpiece with peek inserts (Mini Piezon EMS; PI EMS) .

Different subgroups will be defined according to the material of the dental crown of the related implant.

The mechanical debridement appointments will be carried out at the baseline, after 6 months, and after 12 months, after instruction and motivation of the patient, completion of the clinical chart with the recording of the Probing Depth (evaluation in mm of the peri-implant sulcus taken by a periodontal probe; 4 surfaces of the gingival margin are detected: vestibular, palatal/lingual, mesial, distal), Bleeding on Probing and Plaque Control Record.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70
* Presence of at least one dental implant
* Good compliance

Exclusion Criteria:

* Patients with cardiac stimulators
* Patients with neurological disorders
* Patients with psychological disorders
* Pregnant women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2023-03-30 (Actual); Primary Completion 2025-02-10 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Change in Probing Depth (PD) | Baseline (T0), 6 months (T1), 12 months (T2)
  Evaluation in mm of the peri-implant sulcus taken by a periodontal probe. 4 surfaces of the gingival margin are detected: vestibular, palatal/lingual, mesial, distal.
Change in Bleeding on Probing (BoP) | Baseline (T0), 6 months (T1), 12 months (T2)
  Evaluation of the presence or absence of gingival bleeding during a probing with a dichotomous scoring (yes/no) of bleeding sites. The sum of the bleeding sites is divided for the total sites and multiplied per 100.
Change in Plaque Control Record | Baseline (T0), 6 months (T1), 12 months (T2)
  % assessment of the amount of plaque on dental surfaces; it is detected on 4 surfaces: distal, mesial, vestibular, lingual / palatal. The number of sites with plaque is divided by the total number of sites available in the mouth and multiplied by 100. Results indicate the index as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Scribante, Principal Investigator — University of Pavia
Locations (1):
- Unit of Dental Hygiene - Section of Dentistry - Department of Clinical, Surgical, Diagnostic and Paediatrics - University of Pavia, Pavia, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Data will be available upon motivated request to Principal Investigator.